CLINICAL TRIAL: NCT06353568
Title: Effect of Photobiomodulation as a Preventive Treatment for Diabetic Foot: Randomized Controlled Blinded Clinical Study
Brief Title: Effect of Photobiomodulation as a Preventive Treatment for Diabetic Foot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Kristianne Porta Santos Fernandes, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 5.888.210
Record Dates: First submitted 2024-02-27; First posted 2024-04-09 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Diabetic Foot
Keywords: photobiomodulation; diabetes mellitus; therapeutic education; LED light
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: The PBM Group will use a boot with 1344 LEDs once daily for 6 minutes, over 60 days, and will receive therapeutic education.
  The Control Group will use a non-therapeutic LED boot (placebo) for 6 minutes once daily for 60 days and will also receive therapeutic education.
  Participants will be assessed at the beginning of the study (baseline) and after 30 days (clinical examination) and 60 days (clinical examination, assessment of Peripheral neuropathy, assessment of peripheral artery disease, blood and urine tests, and quality of life evaluation).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: * 1 physician-researcher who will conduct all initial evaluations and follow-up examinations (excluding Doppler ultrasound, Ankle-Brachial Index - ABI, and Toe-Brachial Index - TBI), without knowledge of the subjects' allocation, and will administer the Informed Consent Form (ICF).
  * 1 Vascular surgeon researcher who will perform Doppler ultrasound, Ankle-Brachial Index (ABI), and Toe-Brachial Index (TBI) measurements during the initial assessment and follow-up examinations, without knowledge of the subjects' allocation.
  * 1 Nurse researcher who will retrieve the allocation envelope and provide the appropriate PBM equipment (active or placebo), as well as provide recommendations for its use at home.
  * 1 Researcher, who will not participate in any assessments, will prepare randomization and envelopes to ensure allocation confidentiality.
  * 2 physician residents who will provide daily contact for device usage control, guidance, addressing inquiries, etc.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photobiomodulation Group (Experimental): The PBM Group will use a boot with 1344 LEDs once daily for 6 minutes, over a period of 60 days, and will receive therapeutic education.
  Interventions: Device: Photobiomodulation; Behavioral: Therapeutic education
- Control Group (Sham Comparator): The Control Group will use a non-therapeutic LED boot (placebo) for 6 minutes once daily for 60 days and will also receive therapeutic education.
  Interventions: Device: Simulation of Photobiomodulation; Behavioral: Therapeutic education

INTERVENTIONS:
Device: Photobiomodulation — The PBM Group will use a boot with 1344 LEDs, including 504 LEDs of 660 nm located on the sides of the boot (28.5 mW, 10 J per LED); 504 LEDs of 850 nm also located on the sides of the boot (23 mW, 8 J per LED); 168 LEDs of 660 nm located at the base of the boot (28.5 mW, 10 J per LED); and 168 LEDs of 850 nm also located at the base of the boot (23 mW, 8 J per LED) once daily for 6 minutes, over 60 days.
  Arms: Photobiomodulation Group
Device: Simulation of Photobiomodulation — The Control Group will use a non-therapeutic LED boot (sham procedure) for 6 minutes once daily for 60 days. The boot used is identical to the active boot, but there is no light emission.
  Arms: Control Group
Behavioral: Therapeutic education — Participants will receive therapeutic education regarding nutrition, foot examination, self-care, and guidance on physical activity.

SUMMARY:
This study seeks to evaluate the effect of photobiomodulation (PBM) in the prevention of Diabetic foot (DF), in patients at moderate and high risk for its development, through a controlled, randomized, double-blind clinical trial. Individuals between 18 and 75 years old of both sexes, with type 2 diabetes mellitus (DM), and moderate and high risk for DF will be randomized and allocated into 2 groups of 32 participants each. The PBM Group will use a boot with 1344 LEDs, 504 of which are 660 nm located on the sides of the boot (28.5 milliwatt, 10 J per LED); 504 850 nm also located on the sides of the boot (23 milliwatt, 8 J per LED); 168 of 660 nm located at the base of the boot (28.5 milliwatt, 10 J per LED); 168 of 850 nm also located at the base of the boot (23 milliwatt, 8 J per LED) once a day for 6 minutes, for 60 days and will receive therapeutic education. Participants will be evaluated at baseline, after 30 days (clinical examination) and after 60 days (clinical examination, Peripheral Neuropathy (PN) assessment, Peripheral Artery Disease (PAD) assessment, blood and urine tests, and quality of life).

DETAILED DESCRIPTION:
Diabetic foot (DF) prevention involves risk classification, systemic care, assessment of Peripheral Artery Disease (PAD) and Peripheral Neuropathy (PN), regular foot examination, therapeutic education, and routine use of appropriate footwear. Photobiomodulation (PBM) has been successfully applied in the healing of DF. In addition to the therapeutic effects of PBM, its preventive effects have attracted the attention of researchers. This study seeks to evaluate the effect of PBM in the prevention of DF, in patients at moderate and high risk for its development, through a controlled, randomized, double-blind clinical trial. Individuals between 18 and 75 years old of both sexes, with type 2 DM, and moderate and high risk for DF will be randomized and allocated into 2 groups of 32 participants each. The PBM Group will use a boot with 1344 LEDs, 504 of which are 660 nm located on the sides of the boot (28.5 milliwatt, 10 J per LED); 504 850 nm also located on the sides of the boot (23 milliwatt, 8 J per LED); 168 of 660 nm located at the base of the boot (28.5 milliwatt, 10 J per LED); 168 of 850 nm also located at the base of the boot (23 milliwatt, 8 J per LED) once a day for 6 minutes, for 60 days and will receive therapeutic education. Participants will be evaluated at baseline and after 30 days (clinical examination) and 60 days (clinical examination, PN assessment, PAD assessment, blood and urine tests, and quality of life). The collected data will be stored, and organized in a repository and the appropriate statistical tests will be applied for each specific analysis. In all tests, a significance level of 5% will be adopted.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with type 2 Diabetes Mellitus (according to American Diabetes Association 2021 criteria),
* both sexes,
* between 18 and 75 years,
* Individuals classified, according to the International Working Group on the Diabetic Foot (IWGDF- 2019) scale, as moderate to high risk for developing diabetic foot,

Exclusion Criteria:

* Pregnant women
* Individuals diagnosed with type 1 diabetics,
* Individuals with neuropathy secondary to uncontrolled conditions (hypothyroidism, vitamin B12 deficiency, alcoholism),
* Individuals diagnosed with active infectious condition at the time of inclusion,
* Individuals diagnosed with active ulcer or infectious skin lesion on the legs/feet,
* Individuals with historic of osteomyelitis,
* Individuals with Parkinson's disease,
* Individuals with contracture condition,
* Individuals with severe lower limb ischemia (Fontaine III and IV - Rutherford 4 to 6),
* Individuals with a suspicious skin lesion for neoplasms or cutaneous dysplasias on the legs/feet
* Individuals diagnosed with oncologic disease or undergoing treatment within the last 3 (three) months,
* Individuals presenting unstable angina, recent acute myocardial infarction, history of severe arrhythmia within the last six months,
* Individuals diagnosed with decompensated Chronic Obstructive Pulmonary Disease (COPD),
* Inability to understand the ICF,
* Inability to attend appointments regularly.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-03-30 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Ulcer Incidence | Baseline (Before the intervention)
  The incidence of foot ulcers will be assessed through clinical examination. In addition to these in-person assessments, participants will be monitored daily via telephone contact, during which the researchers (resident physicians) will inquire about any changes in the skin, discomfort, and the use of PBM equipment.
Ulcer Incidence | at 30 days
  The incidence of foot ulcers will be assessed through clinical examination. In addition to these in-person assessments, participants will be monitored daily via telephone contact, during which the researchers (resident physicians) will inquire about any changes in the skin, discomfort, and the use of PBM equipment.
Ulcer Incidence | at 60 days
  The incidence of foot ulcers will be assessed through clinical examination. In addition to these in-person assessments, participants will be monitored daily via telephone contact, during which the researchers (resident physicians) will inquire about any changes in the skin, discomfort, and the use of PBM equipment.

SECONDARY OUTCOMES:
Tactile sensitivity with Semmes-Weinstein monofilament | Baseline (Before the intervention)
  This assessment will be conducted using the Semmes-Weinstein esthesiometer 5.07 with a 10 g filament, following the standard technique outlined in the IWGDF 2019 guidelines, as described in Annex 1. The test will be performed at three different locations on both feet. Protective sensation will be considered present if the patient responds correctly in two out of three applications at each location, and absent if they respond incorrectly in two out of three applications. Each esthesiometer will be used to evaluate a maximum of 10 participants on the same day and discarded after 70 evaluations to maintain accuracy.
Tactile sensitivity with Semmes-Weinstein monofilament | at 60 days
  This assessment will be conducted using the Semmes-Weinstein esthesiometer 5.07 with a 10 g filament, following the standard technique outlined in the IWGDF 2019 guidelines, as described in Annex 1. The test will be performed at three different locations on both feet. Protective sensation will be considered present if the patient responds correctly in two out of three applications at each location, and absent if they respond incorrectly in two out of three applications. Each esthesiometer will be used to evaluate a maximum of 10 participants on the same day and discarded after 70 evaluations to maintain accuracy.
Vibratory sensitivity | Baseline (Before the intervention)
  Participants will be tested with a 128 Hz tuning fork applied to the dorsal aspect of the distal phalanx of the first toe (hallux) or another toe if the hallux is absent. The test will be considered positive if the participant responds correctly to at least two out of three applications and negative if two out of three responses are incorrect
Vibratory sensitivity | at 60 days
  Participants will be tested with a 128 Hz tuning fork applied to the dorsal aspect of the distal phalanx of the first toe (hallux) or another toe if the hallux is absent. The test will be considered positive if the participant responds correctly to at least two out of three applications and negative if two out of three responses are incorrect
Assessment of Achilles reflex | Baseline (Before the intervention)
  The assessment of the Achilles reflex will be conducted with the participant seated, with the foot relaxed and suspended in slight dorsiflexion. A gentle tap will be applied with a reflex hammer to the Achilles tendon. The result will be considered abnormal if plantar flexion reflex of the foot is not observed. The loss of the Achilles tendon reflex is associated with diabetic neuropathy
Assessment of Achilles reflex | at 60 days
  The assessment of the Achilles reflex will be conducted with the participant seated, with the foot relaxed and suspended in slight dorsiflexion. A gentle tap will be applied with a reflex hammer to the Achilles tendon. The result will be considered abnormal if plantar flexion reflex of the foot is not observed. The loss of the Achilles tendon reflex is associated with diabetic neuropathy
Neuropathy Symptom Score (NSS) | Baseline (Before the intervention)
  For the calculation of ESN, patients will be asked about: the sensation of pain or discomfort in the legs and the occurrence, location, timing, and relief of symptoms such as fatigue, cramps, itching, burning, numbness, and tingling in the lower limb. PN will be considered mild when ESN scores between 3 and 4, moderate when between 5 and 6, or severe when reaching 7 to 9 points.
Neuropathy Symptom Score (NSS) | at 60 days
  For the calculation of ESN, patients will be asked about: the sensation of pain or discomfort in the legs and the occurrence, location, timing, and relief of symptoms such as fatigue, cramps, itching, burning, numbness, and tingling in the lower limbs. PN will be considered mild when ESN scores between 3 and 4, moderate when between 5 and 6, or severe when reaching 7 to 9 points.
Neuropathic Impairment Score (NIS) | Baseline (Before the intervention)
  Painful sensitivity will be assessed by applying pressure for 1 second with a blunt-tipped pin on the dorsal surface of the skin near the hallux nail, and thermal sensitivity will be assessed using a metal rod cooled to 32 and 36°C applied at the same location.
  Before the tests, procedures will be demonstrated on the hands. Sensitivities will be scored on each foot as present (0 points) or reduced/absent (1 point). The reflex will be scored as normal (0 points), present with effort (1 point), or absent (2 points). ECN ranges from 0 to 10, obtained by summing the scores of both feet. Values between 3 and 5 indicate mild neuropathy signs, between 6-8 indicate moderate neuropathy signs, and between 9 and 10 indicate severe neuropathy signs
Neuropathic Impairment Score (NIS) | at 60 days
  Painful sensitivity will be assessed by applying pressure for 1 second with a blunt-tipped pin on the dorsal surface of the skin near the hallux nail, and thermal sensitivity will be assessed using a metal rod cooled to 32 and 36°C applied at the same location.
  Before the tests, procedures will be demonstrated on the hands. Sensitivities will be scored on each foot as present (0 points) or reduced/absent (1 point). The reflex will be scored as normal (0 points), present with effort (1 point), or absent (2 points). ECN ranges from 0 to 10, obtained by summing the scores of both feet. Values between 3 and 5 indicate mild neuropathy signs, between 6-8 indicate moderate neuropathy signs, and between 9 and 10 indicate severe neuropathy signs
Evaluation of the degree of ischemia | Baseline (Before the intervention)
  The ankle-brachial index (ABI) will be measured by placing the sphygmomanometer cuff in the usual manner on the UL (above the elbow crease) and just above the ankle bones (ankle) on the LL with the patient in a supine position; inflating the cuff until the sound of blood flow becomes inaudible and then deflating it until the first sound of blood flow is heard, which corresponds to the maximum systolic pressure. Measurements will be repeated three times.
Evaluation of the degree of ischemia | at 60 days
  The ankle-brachial index (ABI) will be measured by placing the sphygmomanometer cuff in the usual manner on the UL (above the elbow crease) and just above the ankle bones (ankle) on the LL with the patient in a supine position; inflating the cuff until the sound of blood flow becomes inaudible and then deflating it until the first sound of blood flow is heard, which corresponds to the maximum systolic pressure. Measurements will be repeated three times.
Systolic peak velocity | Baseline (Before the intervention)
  In the distal segments of the anterior and posterior tibial arteries and fibular artery in cm²/s measured by Doppler ultrasound.
Systolic peak velocity | at 60 days
  In the distal segments of the anterior and posterior tibial arteries and fibular artery in cm²/s measured by Doppler ultrasound.
Resistance Index | Baseline (Before the intervention)
  In the distal segments of the anterior and posterior tibial arteries and fibular artery - calculated by the formula (systolic peak velocity - diastolic peak velocity) / systolic peak velocity.
Resistance Index | at 60 days
  In the distal segments of the anterior and posterior tibial arteries and fibular artery - calculated by the formula (systolic peak velocity - diastolic peak velocity) / systolic peak velocity.
Waveform pattern | Baseline (Before the intervention)
  The waveform pattern of the distal segments of the anterior and posterior tibial arteries and fibular artery in Doppler ultrasound examination will be classified as triphasic, biphasic, or monophasic.
Waveform pattern | at 60 days
  The waveform pattern of the distal segments of the anterior and posterior tibial arteries and fibular artery in Doppler ultrasound examination will be classified as triphasic, biphasic, or monophasic.
Evaluation of claudication | Baseline (Before the intervention)
  The accuracy of using the Edinburgh Claudication Questionnaire alone is debatable, but this instrument can be used as a complement to clinical evaluation data for PAD. The questionnaire consists of 6 questions and has been validated for Portuguese. The definition of positive claudication requires the following set of responses: 1 = "yes", 2 = "no", 3 = "yes", 5 = "usually disappears in 10 minutes or less", and 6 = "calf" and/or "thigh" and/or "buttock" (regardless of whether other locations are marked) or NEGATIVE if any different combination is marked. Question 4 is not used to define the presence but rather the severity of claudication: "No" = Grade 1 (mild severity); and "Yes" = Grade 2.
Evaluation of claudication | at 60 days
  The accuracy of using the Edinburgh Claudication Questionnaire alone is debatable, but this instrument can be used as a complement to clinical evaluation data for PAD. The questionnaire consists of 6 questions and has been validated for Portuguese. The definition of positive claudication requires the following set of responses: 1 = "yes", 2 = "no", 3 = "yes", 5 = "usually disappears in 10 minutes or less", and 6 = "calf" and/or "thigh" and/or "buttock" (regardless of whether other locations are marked) or NEGATIVE if any different combination is marked. Question 4 is not used to define the presence but rather the severity of claudication: "No" = Grade 1 (mild severity); and "Yes" = Grade 2.
Thermography | Baseline (Before the intervention)
  . To utilize this technique, the imaging room should be climate-controlled with a stabilized temperature between 21 and 23°C. After removing shoes and socks, participants will lie in a supine position with a pillow under their legs without ankle support, keeping their legs slightly apart for at least 15 minutes to allow temperature equilibrium and circulation stabilization of the limbs. Participants will be instructed to clean their lower limbs or take a bath at least 2 hours before the examination, avoid physical activity on the day of the examination, and refrain from applying creams or any substances to the lower limbs. Infrared images (thermograms) will be captured by a highly sensitive infrared sensor (18mm, resolution 320x240 pixels), Flir T420®, supported on a tripod maintained at 150 cm from the participants' foot soles, and a 15 cm ruler will be included in each image.
Thermography | at 60 days
  . To utilize this technique, the imaging room should be climate-controlled with a stabilized temperature between 21 and 23°C. After removing shoes and socks, participants will lie in a supine position with a pillow under their legs without ankle support, keeping their legs slightly apart for at least 15 minutes to allow temperature equilibrium and circulation stabilization of the limbs. Participants will be instructed to clean their lower limbs or take a bath at least 2 hours before the examination, avoid physical activity on the day of the examination, and refrain from applying creams or any substances to the lower limbs. Infrared images (thermograms) will be captured by a highly sensitive infrared sensor (18mm, resolution 320x240 pixels), Flir T420®, supported on a tripod maintained at 150 cm from the participants' foot soles, and a 15 cm ruler will be included in each image..
Quality of Life Assessment | Baseline (Before the intervention)
  The quality of life of individuals will be assessed using the Diabetes-21 instrument, which is a multidimensional scale adapted from the Diabetes-39, validated for Brazilian Portuguese.
Quality of Life Assessment | at 60 days
  The quality of life of individuals will be assessed using the Diabetes-21 instrument, which is a multidimensional scale adapted from the Diabetes-39, validated for Brazilian Portuguese.

CONTACTS AND LOCATIONS:
Overall Officials: Kristianne KS Fernandes, PhD, Principal Investigator — University of Nove de Julho
Locations (1):
- Conjunto Hospitalar do Mandaqui, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Lourenco R, Perez ST, Motta LJ, Duran CCG, Padilha ARS, Bussadori SK, Malavazzi TCDS, Horliana ACRT, Mesquita-Ferrari RA, Fernandes KPS. Effect of photobiomodulation as preventive treatment of diabetic foot ulcer: randomised, controlled, double-blind, clinical trial protocol. BMJ Open. 2025 Jan 22;15(1):e094594. doi: 10.1136/bmjopen-2024-094594. PMID 39843368